CLINICAL TRIAL: NCT02385526
Title: ASCEND: Vagus Nerve Stimulation Titration Protocol to Improve Tolerance and Accelerate Adaptation
Brief Title: Vagus Nerve Stimulation Titration Protocol to Improve Tolerance and Accelerate Adaptation
Acronym: ASCEND
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Organization: LivaNova (Industry)
Other Study IDs: E-40
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-10

CONDITIONS: Epilepsy; Seizures
Keywords: Vagus Nerve Stimulation; ASCEND; VNS Titration to Improve Tolerance and Accelerate Adaptation
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Vagus Nerve Stimulation Therapy Standard Titration
  Interventions: Device: Vagus Nerve Stimulation Therapy
- Group B: Vagus Nerve Stimulation Therapy Alternate Titration 1
  Interventions: Device: Vagus Nerve Stimulation Therapy
- Group C: Vagus Nerve Stimulation Therapy Alternate Titration 2
  Interventions: Device: Vagus Nerve Stimulation Therapy

INTERVENTIONS:
Device: Vagus Nerve Stimulation Therapy — Stimulation of the left tenth cranial nerve via VNS Therapy
  Other Names: VNS Therapy

SUMMARY:
Post-market, on-label, double-blind, randomized, prospective, interventional, tolerability and clinical outcomes study to determine the number of patients achieving their final assigned VNS Therapy dose settings in patients with drug-resistant epilepsy who are being treated with adjunctive VNS Therapy using new titration protocols.

DETAILED DESCRIPTION:
Post-market, on-label, double-blind, randomized, prospective, interventional, tolerability and clinical outcomes study is designed to determine which VNS Therapy titration paradigm allows more patients to achieve a therapeutic dose within a specified time frame. Additionally, the study will collect data on the acute tolerability and clinical outcomes for patients with drug-resistant epilepsy treated with adjunctive VNS Therapy employing three different titration paradigms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must agree to be treated with VNS Therapy. The decision to treat with VNS Therapy must have been made independent of and prior to participation in the study.
2. Patients must be 12 years or older and have partial onset seizures or must follow the indication for use statement for VNS Therapy.
3. Patient and/or caregiver must be able and willing to give accurate side effect reports, global impressions data and complete study instruments with minimal assistance throughout the study.
4. Patient or legal guardian understands study procedures and voluntarily signs an informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional policies. In the event the patient is under the age of 18, the patient will also be required to sign an assent affirming agreement to participate in research according to local IRB requirements.
5. Patient must be taking at least 1 anti-epileptic drug treatment

Exclusion Criteria:

1. Patient currently uses, or is expected to use during the study, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy.
2. Patient is expected to require MRI using a body coil for transmission of RF during the clinical study.
3. Patient has a progressive neurological condition (e.g. brain tumor etc.).
4. In the investigator's opinion, the patient or legal guardian is unable to comply with the frequency of clinic visits during the study.
5. Patient is currently using an investigational device or pharmacologic medication not approved by the FDA.
6. Patient was previously implanted with VNS Therapy.
7. In the investigator's opinion, the patient is considered a suicide risk or is otherwise not a good candidate for this study.
8. Patient/Caregiver is unable to complete the required study follow-up visits and assessments.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study shall include adults and adolescents over 12 years of age with partial onset seizures that are refractory to antiepileptic medications and eligible for VNS Therapy indicated for use as an adjunctive therapy in reducing the frequency of seizures.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Way, Study Director — Cyberonics, Inc.
Locations (15):
- United States (15):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Loma Linda University, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St. Joseph's Hospital, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Mercy Medical Research Institue, Springfield, Missouri
  - University of Nebraska, Omaha, Nebraska
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Covenant Hospital, Lubbock, Texas
  - Scott & White Healthcare, Temple, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Bagic AI, Verner R, Afra P, Benbadis S; ASCEND Study Group. ASCEND: A randomized controlled trial of titration strategies for vagus nerve stimulation in drug-resistant epilepsy. Epilepsy Behav. 2023 Aug;145:109333. doi: 10.1016/j.yebeh.2023.109333. Epub 2023 Jul 8. PMID 37429122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled at 15 clinical sites including university and private hospital clinics. Enrollment was allowed following successful initiation of the first clinical site on 04MAR2015 and closed on 29JUN2016. The first subject enrolled on 28APR2015 and the final two subjects enrolled on 29JUN2016. The final subject exited the study on 10OCT2016.
Pre-assignment Details: All subjects were required to receive implantation of a commercially available Vagus Nerve Stimulation generator (Stimulation of the left tenth cranial nerve via VNS Therapy) prior to randomization. The generator was to remain "off" until after randomization completion.
Groups:
- Group A: Vagus Nerve Stimulation Therapy Standard Titration method
- Group B: Vagus Nerve Stimulation Therapy Alternate Titration 1
  Alternate titration method that combined methods from Group A and Group C.
- Group C: Vagus Nerve Stimulation Therapy Alternate Titration 2
  Alternate titration method used in the ANTHEM-HF trial which evaluated the performance of autonomic regulation using VNS Therapy in patients with chronic symptomatic heart failure and reduced ejection fraction.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 22 | 20 | 20
Completed | 20 | 17 | 20
Not Completed | 2 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 22 | 20 | 20 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 21 | 19 | 19 | 59
  >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 10 | 37
  Male | 6 | 9 | 10 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Non-Hispanic | 15 | 17 | 13 | 45
  Race/Ethnicity: Black or African American | 3 | 1 | 1 | 5
  Race/Ethnicity: Hispanic or Latino | 4 | 2 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 20 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percent Patients Reaching the Defined Target Dose
Description: Determination of the proportion (percent) of patients in each VNS Therapy titration group reaching the defined target dose within clinically defined titration time-frame
Time Frame: 12 weeks post implant
Population: Population of subjects implanted with Vagus Nerve Therapy generator who received stimulation via left, tenth cranial nerve at varying dosing methods (device settings adjustments) depending on the group each subject was randomized. All subject had a common, final target dose to achieve but used alternate methods to achieve the target dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 22 | 20 | 20
Participants | 18 | 9 | 12

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of each subjects study participation of 12 weeks. This period began from the first enrollment 28APR2015 to the final exit 10OCT2016.
Description: Adverse reporting occurred via subject reporting and investigator assessment during the scheduled subject visits. Events related to epilepsy were not to be recorded unless a worsening from baseline was observed or experienced.
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 9/22 | 7/20 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=22) | Group B (N=20) | Group C (N=20)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Peripheral vascular disease of right superficial femoral artery (Post Implant) unrelated to implant or stimulation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=22) | Group B (N=20) | Group C (N=20)
Palpatations [S] (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Cerumen impaction [U] (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Tinnitus [U] (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Constipation [U] (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Diarrhoea [U] (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Dysphagia [S] (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Chest Pain [S] (General disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Discomfort [S] (General disorders) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Fatigue [S] (General disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Implant site hoematoma [I] (General disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Medical device discomfort [S] (General disorders) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Medical device pain [S] [SI] (General disorders) | 1 (1) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Non-cardiac chest pain [S] (General disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Cellulitis [U] (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Lower respiratory tract infection [U] (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Nasopharyngitis [U] (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Staphyloccal infection [I] (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Urinary tract infection [U] (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Incision site haematoma [U] (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Incision site hypoaesthesia [I] (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Incision site pain [I] (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Post procedural haemorrhage [U] (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Procedural headache [S] (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Procedural nausea [U] (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Arthralgia [U] (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Back pain [U] (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Muscle spasms [S] (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Muscle tightness [SI] (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Muscle twitching [S] (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Myalgia [I] (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Neck pain [I] (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Pain in extremety [I] (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Pain in jaw [U] [S] (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Convulsion [U] (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Headache [U] (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Migraine [U] (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Paraesthesia [S] (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Postural tremor [S] (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Somnolence [U] (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Anxiety [U] [SI] (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Asthma [U] (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Cough [S] (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Dysphonia [S] (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Oropharyngeal pain [I] [S] (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Sleep apnoea syndrome [S] (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Sputum increased [SI] (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Throat tightness [S] (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Pruritis [S] (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant
Peripheral arterial occlusive disease [U] (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) — [S] Related to Stimulation [I] Related to Implant [SI] Related to Stimulation and Implant [U] Unrelated to Stimulation or Implant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days